CLINICAL TRIAL: NCT00497757
Title: 1) Induction of Donor-Specific Tolerance in Recipients of Cardiac Allografts by Donor Stem Cell Infusion 2) Induction of Donor-Specific Tolerance by Donor Facilitating Cell (FC): Stem Cell Infusion in Recipients of Hepatic Allografts
Brief Title: Induction of Donor Specific Tolerance in Recipients of Cardiac Allografts by Donor Stem Cell Infusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzanne T. Ildstad (Other)
Responsible Party: Sponsor-Investigator, Suzanne T. Ildstad, Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT-7494-041698
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Heart Transplantation
Keywords: Marrow/hematopoietic stem cell transplant

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cardiac Failure Patients (Experimental): Recipients treated with an enriched hematopoetic stem cell infusion from the heart donor's bone marrow
  Interventions: Biological: enriched hematopoetic stem cell infusion

INTERVENTIONS:
Biological: enriched hematopoetic stem cell infusion — Enriched Hematopoetic Stem Cell Infusion

SUMMARY:
The goal of this research study is to establish chimerism and avoid graft-versus-host disease in patients who need a heart transplant.

DETAILED DESCRIPTION:
At the present time, heart transplant recipients must take anti-rejection medication to prevent rejection of the donated heart. Even with this medication, chronic rejection is the most common cause of late graft loss. The anti-rejection agents themselves are significantly toxic, with side effects including kidney damage, infection and an increased incidence of cancer. The goal of this study is to allow the patient to develop "tolerance" to the transplanted heart while maintaining a competent immune system. Tolerance enables the transplant recipient's body to recognize the transplanted organ as self rather than foreign tissue. The recipient will not try to reject the donor heart and the need for anti-rejection medication could be dramatically decreased or eliminated entirely. To accomplish this, patients in this study will receive specially treated bone marrow taken from their heart donor. Bone marrow transplant has been shown in animal studies and in humans to induce tolerance following organ transplant.

Two factors limit the application of donor marrow transplant to induce tolerance: 1) preparing the patient for transplant (conditioning); and 2) graft-versus-host disease (GVHD). Traditional conditioning destroys the recipient's immune system and requires that the marrow transplant be successful because the patient is unable to fight off infection if the donor cells do not survive. GVHD occurs when donor immune cells recognize the recipient's cells as foreign tissue and attack them. Severe GVHD can result in death. This study utilizes a new approach to conditioning which leaves the patient's immune system intact. The transplant product is depleted of GVHD-producing cells but retains tolerance-promoting facilitating cells, which are intended to ensure the donor and recipient cells coexists peacefully, a state called mixed chimerism. The toxicity of conditioning and transplantation is significantly reduced.

In this study, we will determine the appropriate cell dose to safely establish mixed chimerism following partial conditioning in heart transplant recipients. The study takes a gradual approach to increasing the cell dose to achieve mixed chimerism. We believe this study will provide a breakthrough in the approach to heart transplantation. Our goal is to evaluate the potential of safely establishing mixed chimerism to induce tolerance following heart transplant and reduce or eliminate the need for anti-rejection therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between the ages of 18 and 70 years and meet the institution's criteria for cardiac transplantation.
* Subjects must have acceptable negative results for infectious disease markers done within two weeks of the bone marrow infusion.
* Subject is receiving a first cardiac transplant.
* Subjects receiving a multi-organ transplant (i.e., heart/kidney) may be included at the discretion of the PI and investigators.

Note: These multi-organ subjects will have identical criteria with the exception of adequate function of the affected organ to be transplanted (i.e., kidney). They are included in the total of thirty subjects to be transplanted.

* Subject's panel reactive antibody (PRA) is <40. If the patient is plasmapheresed prior to the heart transplant, then the pre-transplant PRA will not be a consideration for inclusion/exclusion.
* Subject must have a negative crossmatch with the donor.
* Women who are of child bearing potential must have a negative pregnancy test (urine test within 48 hours) before TBI and agree to use reliable contraception for one year following transplant.
* Subject is able to give informed consent.

Exclusion Criteria:

* Clinically active bacterial, fungal, viral or parasitic infection
* Pregnancy
* Previous radiation therapy at a dose that would preclude TBI
* Subject is unable to give informed consent
* If the procedures associated with the study (i.e., delivering TBI) would significantly extend the cold ischemia time of the heart, the protocol will be abandoned and the patient will receive a conventional heart transplant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-07; Primary Completion 2011-11-07 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Enriched Hematopoetic Stem Cell Engraftment | One month to three years

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne T Ildstad, MD, Study Director — University of Louisville

IPD SHARING:
Plan to Share IPD: No